CLINICAL TRIAL: NCT01968044
Title: A Multicenter,Randomized, Placebo-controlled, Parallel Group, Double-blind, Phase IIIb Study to Evaluate the Safety and Efficacy After 12 Weeks Administration of Gemigliptin and Placebo in Type 2 Diabetes Mellitus Patients With Moderate or Severe Renal Impairment With an Additional 40 Weeks, Double-blind,Active-controlled, Double-dummy,Long-term Extension Study
Brief Title: A Phase IIIb Study to Evaluate the Safety and Efficacy of Gemigliptin in Type 2 Diabetes Mellitus Patients With Moderate or Severe Renal Impairment(GUARD Study)
Acronym: GUARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-DPCL015
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 DM Patients With Moderate or Severe Renal Impairment
Keywords: renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Gemigliptin (Experimental): Participant will remain gemigliptin 50mg throughout entire study (52 weeks).
  Interventions: Drug: Gemigliptin
- Placebo to linagliptin (Other): Participant who is randomized to placebo will be switched to linagliptin after 12 week and administered linagliptin by week 52.
  Interventions: Drug: Placebo to Linagliptin

INTERVENTIONS:
Drug: Gemigliptin
  Arms: Gemigliptin
Drug: Placebo to Linagliptin
  Arms: Placebo to linagliptin

SUMMARY:
Therapuetic options are limited for Type 2 Diabetes Mellitus (T2DM) pateints with renal impairment. This clinical study is to asses safety and efficacy of the DPP-4 inhibitor gemigliptin in patients with type 2 DM and moderate or severe renal impairment for long-term peirod (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus
* Patients with moderate or severe renal insufficiency
* All patients give written informed consent

Exclusion Criteria:

* Has type 1 diabetes mellitus or a history of ketoacidosis
* Is on dialysis or is likely to need dialysis during the study
* Has active liver disease

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
HbA1c change | HbA1c change from baseline to week 12

SECONDARY OUTCOMES:
HbA1c Change | HbA1c change from baselint to week 6, 52
FPG | FPG change from baseline to week 6,12,52
Glycated albumin | Glycated albumin change from baseline to week 6,12,52
Fructosamin | Fructosamin change from baseline to week 6,12,52
Waist | Waist change from baseline to week 12,52
HbA1c responser (HbA1c<7.0%) | HbA1c responser rate at week 12,52
Fasting serum C-peptide | Fasting serum C-peptide change from baseline to week 12,52
Fasting Lipid parameters | Fasting Lipid parameters change from baseline to week 12,52
Albuminuria | Albuminuria change from baseline to week 12,52

CONTACTS AND LOCATIONS:
Overall Officials: DR Cha, MD, Ph.D, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Seoul, South Korea